CLINICAL TRIAL: NCT01292538
Title: A Double-blind, Placebo-controlled Randomized Evaluation of the Effect of the Erchonia Scanner Device (GLS) Green Diode on Body Contouring of the Waist, Hips and Thighs
Brief Title: Study of the Effectiveness of Green Diode Laser Light on Body Shaping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC-GREEN001
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Body Contouring

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia GLS 532nm (Experimental): 532nm green laser light therapy.
  Interventions: Device: Erchonia GLS
- Placebo laser (Sham Comparator): Sham light output with no therapeutic benefit
  Interventions: Device: Placebo laser

INTERVENTIONS:
Device: Erchonia GLS — 532 nm green diode low level laser light device
  Arms: Erchonia GLS 532nm
Device: Placebo laser — Sham light output with no therapeutic benefit
  Arms: Placebo laser

SUMMARY:
The purpose of this study is to determine if 532nm green diode laser light is effective in body contouring of the waist, hips and thighs.

DETAILED DESCRIPTION:
Weight loss and body contouring are large, constantly-growing fields of cosmetic surgery. However, while the demand for body shaping procedures is constantly on the rise, so is the demand for such procedures to be performed more quickly, simply and most importantly, less invasively; hence the growing popularity of non- to minimally-invasive cosmetic surgery procedures. In 2005, more than 7.5 million minimally-invasive cosmetic procedures were performed, a 35% increase from 2000.

In recent years, Erchonia Corporation, a manufacturer of low level lasers, has developed a dual-diode laser that emits 532 nm and 635nm collimated line-generated beams to emulsify fat. In August, 2010, the Erchonia® ML Scanner (MLS) 635nm was cleared by FDA for use as a non-invasive dermatological aesthetic treatment for the reduction of circumference of hips, waist, and thighs. It was determined that the biochemical effect of the Erchonia® MLS stimulates the mitochondria of the adipocyte cells which in turn increases the production of ATP. The newly synthesized ATP triggers the up-regulation of cyclic adenosine monophosphate (cAMP). cAMP has been shown to stimulate cytoplasmic lipase, triggering the conversion of triglycerides into fatty acids and glycerol that can easily pass through the cell membrane. The transitory pore is evidence that the laser is allowing for the movement of fatty acids, glycerol, and triglycerides to pass across the membrane and into extra-cellular space. Through vasodilation of nearby blood vessels and arteries, oxidization of the triglycerides and fatty acids occurs within the extra-cellular space.

This pilot study will apply the Erchonia® MLS employing 532 nm green diodes in lieu of 635 nm red diodes to compare the results to those attained using the 635 nm diodes. The Sponsor believes the use of 532 nm diodes may prove as effective as 635 nm diodes combined with a reduction in total procedure administration time from 40 to 30 minutes. It is the goal of this study to evaluate this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) less than 30 kg/m²
* Subject indicated for liposuction or use of liposuction techniques for the removal of localized deposits of adipose tissues that do not respond to diet and exercise; specifically for the indication of body contouring in the areas of the waist, hips and bilateral thighs. (As per the American Academy of Cosmetic Surgery's 2006 Guidelines for Liposuction Surgery).
* Subject is willing and able to abstain from partaking in any treatment other than the study procedure to promote body contouring and/or weight loss during study participation.
* Subject is willing and able to maintain his or her regular diet and exercise regimen without effecting significant change in either direction during study participation.

Exclusion Criteria:

* Body Mass Index (BMI) of 30 kg/m² or greater.
* Diabetic dependent on insulin or oral hypoglycemic medications.
* Known cardiovascular disease.
* Prior cardiac surgery.
* Prior surgical intervention for body sculpting/weight loss, such as liposuction, abdominoplasty, stomach stapling, lap band surgery.
* Medical, physical, or other contraindications for body sculpting/weight loss.
* Use of medication(s) known to affect weight levels and/or to cause bloating or swelling and for which abstinence during study participation is not safe or medically prudent.
* Any medical condition known to affect weight levels and/or cause bloating or swelling.
* Diagnosis of, and/or taking medication for, irritable bowel syndrome.
* Active infection, wound or other external trauma to the areas to be treated with the laser.
* Photosensitivity disorder.
* Current cancer or receiving treatment for cancer.
* Pregnant, breast feeding, or planning pregnancy prior to study end.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to record study measurements.
* Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to weight-related/body shape issues.
* Participation in research in the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Roche, MD, FACS, Principal Investigator; Robert F Jackson, MD, FACS, Principal Investigator
Locations (2):
- United States (2):
  - Surgeon's Inc., Marion, Indiana
  - Bloomfield Laser and Cosmetic Surgery Center, Bloomfield Hills, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia GLS 532nm | Placebo Laser
Started | 35 | 32
Completed | 35 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia GLS 532nm | Placebo Laser | Total
Number analyzed (Participants) | 35 | 32 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.60 (10.05) | 39.03 (10.16) | 38.04 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 32 | 61
  Unknown or Not Reported | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Combined Circumference in Inches of the Waist, Hips and Bilateral Thighs
Description: Mean change in total combined circumference inches of the waist, hips and bilateral thighs from baseline to endpoint evaluation.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Erchonia GLS 532nm | Placebo Laser
Number analyzed (Participants) | 35 | 32
inches | -3.895 (3.03) | -1.136 (2.27)

ADVERSE EVENTS:
Arm/Group | Erchonia GLS 532nm | Placebo Laser
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32
Other Adverse Events (participants affected / at risk) | 0/35 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No